CLINICAL TRIAL: NCT00476736
Title: Reassessment Study of The Effect of N-Acetylcystein on Quality of Life and Air Trapping During Rest and After Exercise
Brief Title: The Effect of N-Acetylcystein on Quality of Life and Air Trapping During Rest and After Exercise
Acronym: NAC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 56/07
Record Dates: First submitted 2007-05-21; First posted 2007-05-22 (Estimated); Last update posted 2007-05-22 (Estimated); Status verified 2007-05

CONDITIONS: Quality of Life; Exercise
Keywords: COPD; Pulmonary function; Air trapping; Acetyl cystein
MeSH Terms: conditions — Motor Activity; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Effect on small airways (N-Acetylcystein)

SUMMARY:
Treatment of COPD patients depends on the stage of the disease. First of all it is strongly recommended quit smoking, then bronchodilators drugs are added. In more advanced stages inhaled corticosteroids and pulmonary rehabilitation are added. In hypoxemic patients a long term supplemental oxygen is advised.

The addition of sputum modifiers drugs is equivocal, since no objective improvement was documented.

N-Acetylcystein (NAC) is a drug known for its anti-oxidant and mucolytic activity. In animal models of disease it showed its beneficial activity , whereas in human such changes weren't demonstrated. In all the studies FEV1 was used to demonstrate the beneficial effect of the drug, although the disease changes are at the level of small airways which is almost not expressed by the measurement FEV1.

Purpose of the study

1. To estimate the damage severity at the small airways.
2. To estimate the change in quality of life.
3. To assess the pulmonary function changes at rest and following exercise, including parameters of air trapping (hyperinflation)

Methods & Materials Patients - Inclusion - 30 Moderate COPD (GOLD classification) , AGE 45-70, both sexes. Treated with inhaled steroids and long acting beta agonists.

Exclusion - Active ischemic heart disease, heart failure, orthopedic problems that preclude ergometric bicycle activity.

Questionnaire - The St. George questionnaire for quality of life will be used . Pulmonary function testing- Lung volumes and spirometry un including inspiratory capacity will be measured before and after exercise.

Study protocol - 2 weeks run in, for observation disease stability and drug adherence.

Patient will randomly separated in 2 groups . Group A - will receive 600-1200 mg N-acetyl cystein twice daily. Group B - will receive as control placebo . Following 4 weeks of treatment patient will clinically re-examined and PFT's performed as described. After 2 weeks of washout group A. will serve as control and group B. will be treated with NAC as described.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a major cause of chronic morbidity and mortality throughout the world. Many people suffer from this disease for years and die prematurely from it or its complications. COPD is the fourth leading cause of death in the world, and further increases in its prevalence and mortality can be predicted in the coming decades. COPD is characterized by a slowly progressing, irreversible airflow limitation caused by chronic inflammation in the bronchioles. It is diagnosed by performing spirometry. In the early stages, COPD can be asymptomatic, although episodes of coughing, often with sputum production, are not rare. In more advance stages, when there are also symptoms of shortness breath on exertion, a significant part of lung function may be reduced. The diagnosis of COPD is usually established in the later stages, and this diagnostic delay may either be due to the patient's gradual adaptation to a decreasing lung function or denial of the disease. In addition, because doctors are unaware of, or not responding to the symptoms of the patient. The main cause of COPD is smoking and it often manifests itself after someone has been smoking more than 20 cigarettes a day over 20 years (20 pack years). A smoker who is "sensitive" to cigarette smoke may therefore have spirometric changes between the ages of 40 to 45 years if they started smoking as a teenager or early 20th. It has been estimated that 15-20% of smokers develop COPD, but more recent research suggests that as many as 50% develop COPD if the smoker reaches a high age.

Treatment of COPD patients depends on the stage of the disease. First of all it is strongly recommended quit smoking, then bronchodilators drugs are added. In more advanced stages in inhaled corticosteroids and pulmonary rehabilitation are added. In hypoxemic patients a long term supplemental oxygen is advised.

The addition of sputum modifiers drugs is equivocal, since no objective improvement was documented.

N-Acetylcystein (NAC) is a drug known for its anti-oxidant and mucolytic activity. In animal models of disease it showed its beneficial activity , whereas in human such changes weren't demonstrated. In all the studies FEV1 was used to demonstrate the beneficial effect of the drug, although the disease changes are at the level of small airways which is almost not expressed by the measurement FEV1.

Purpose of the study

1. To estimate the damage severity at the small airways.
2. To estimate the change in quality of life.
3. To assess the pulmonary function changes at rest and following exercise, including parameters of air trapping (hyperinflation)

Methods & Materials Patients - Inclusion - 30 Moderate COPD (GOLD classification) , AGE 45-70, both sexes. Treated with inhaled steroids and long acting beta agonists.

Exclusion - Active ischemic heart disease, heart failure, orthopedic problems that preclude ergometric bicycle activity.

Questionnaire - The St. George questionnaire for quality of life will be used . Pulmonary function testing- Lung volumes and spirometry un including inspiratory capacity will be measured before and after exercise.

Study protocol - 2 weeks run in, for observation disease stability and drug adherence.

Patient will randomly separated in 2 groups . Group A - will receive 600-1200 mg N-acetyl cystein twice daily. Group B - will receive as control placebo . Following 4 weeks of treatment patient will clinically re-examined and PFT's performed as described. After 2 weeks of washout group A. will serve as control and group B. will be treated with NAC as described.

ELIGIBILITY:
Inclusion Criteria:

* 30 Moderate COPD (GOLD classification) , AGE 45-70, both sexes.
* Treated with inhaled steroids and long acting beta agonists.

Exclusion Criteria:

* Active ischemic heart disease, heart failure, orthopedic problems that preclude ergometric bicycle activity.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-05; Study Completion 2007-05 (Estimated)

PRIMARY OUTCOMES:
inspiratory capacity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David Stav, Study Chair — Tel Aviv University
Locations (1):
- Pulmonary Institute, Assaf Harofeh Medical Center, Beer Yaakov, Israel

REFERENCES:
- [Derived] Stav D, Raz M. Effect of N-acetylcysteine on air trapping in COPD: a randomized placebo-controlled study. Chest. 2009 Aug;136(2):381-386. doi: 10.1378/chest.09-0421. Epub 2009 May 15. PMID 19447919